CLINICAL TRIAL: NCT00219115
Title: A 12-week Randomized Double-blind Parallel Group Study to Evaluate the Efficacy and Safety of the Combination Aliskiren With HCTZ Compared to Irbesartan or Amlodipine With HCTZ or HCTZ Alone in Hypertensive Patients With BMI ≥ 30 kg/m2 Not Adequately Responsive to HCTZ 25 mg
Brief Title: A Clinical Study to Compare Combination of Aliskiren+ HCTZ to Irbesartan+ HCTZ or Amlodipine+ HCTZ or HCTZ Alone in Obese Hypertensive Not Responsive to HCTZ 25 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2309
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, irbesartan, amlodipine, hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To evaluate the blood pressure lowering effects of the combination of aliskiren 300 mg and HCTZ 25 mg in obese patients with essential hypertension inadequately treated with HCTZ 25 mg, compared to irbesartan or amlodipine with HCTZ or HCTZ alone.

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients with body mass index ≥ 30 kg/m2

Exclusion Criteria

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of Hypertensive encephalopathy or cerebrovascular accident.

Other protocol-defined inclusion exclusion criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2005-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure after 8 weeks
Evaluate number mean sitting systolic/diastolic response from baseline to weeks 4 and 8
Mean sitting diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after week 8
Achieve mean sitting blood pressure control target of < 140/90 mmHg after week 8

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Result] Jordan J, Engeli S, Boye SW, Le Breton S, Keefe DL. Direct Renin inhibition with aliskiren in obese patients with arterial hypertension. Hypertension. 2007 May;49(5):1047-55. doi: 10.1161/HYPERTENSIONAHA.106.084301. Epub 2007 Mar 12. PMID 17353513